CLINICAL TRIAL: NCT04998032
Title: Efficacy and Safety of Once-weekly Supaglutide Versus Placebo in Patients With Type 2 Diabetes Suboptimally Controlled on Metformin: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: A Study of Efficacy and Safety of Supaglutide in Type 2 Diabetes Patients On Metformin Treatment(SUPER-2)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Yinnuo Pharmaceutical Technology Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YN011-302
Record Dates: First submitted 2021-07-28; First posted 2021-08-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: This clinical trial includes dosage determination (Phase IIb) and efficacy confirmation stage(Phase III ). During the phase IIb, subjects were randomly assigned to Supaglutide 1mg + metformin, Supaglutide 3mg + metformin and placebo + metformin according to a 1:1:1 ratio.
  When 120 subjects complete the 12 weeks of follow-up, Interim analysis will be performed and the results be evaluated by IDMC to confirm the RP3D dose.
  And then during the phase III, subjects were randomly assigned to Supaglutide RP3D + metformin, placebo + metformin group according to a 1:1 ratio.
Who Masked: Participant, Investigator
Masking Description: This includes a 24-week double-blind treatment period, followed by a 28-week open-label treatment period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supaglutide RP3D dose+metformin (Experimental): Supaglutide Subcutaneous injection once a week for 52weeks,combined with metformin
  Interventions: Biological: supaglutide injection+metformin
- placebo+metformin (Placebo Comparator): Placebo Subcutaneous injection once a week for 52weeks,,combined with metformin
  Interventions: Other: placebo+metformin

INTERVENTIONS:
Biological: supaglutide injection+metformin — supaglutide subcutaneous injection under RP3D dose combined with metformin treatment
  Arms: supaglutide RP3D dose+metformin
Other: placebo+metformin — placebo subcutaneous injection combined with metformin treatment
  Arms: placebo+metformin

SUMMARY:
This is a study to evaluate the efficacy and safety of Supaglutide injection in the treatment of type 2 diabetes patients with poor glycemic control after metformin treatment.

This trial includes dosage determination (Phase IIb) and efficacy confirmation stage(Phase III ). The primary outcome of the phase IIb period is to preliminarily evaluate the efficacy and safety of Supaglutide combined with metformin and to provide the recommended dosage for the Phase 3 period after 12-week treatment.

The primary outcome of the Phase III period is to evaluate the efficacy and safety of Supaglutide combined with metformin treatment after 24-week, double-blind treatment. The secondary outcome is to evaluate the efficacy and safety of Supaglutide combined with metformin during the 24-week, double-blinded plus 28-week, open-label treatment period.

DETAILED DESCRIPTION:
This trial includes a 2-week screening period, a 4-week metformin titration and dose-stabilization period, a 4-week induction period, a 24-week double-blind treatment period and a 28-week open-label treatment period, followed by a 4-week follow-up period and a follow-up visit. We calculated that the sample size would need to be 632, including 120 subjects in the period of Phase IIb and 512 subjects in the period of Phase III. During the phase IIb period, subjects were randomly assigned to once-weekly subcutaneously injected Supaglutide 1mg plus metformin, 3mg plus metformin and placebo plus metformin at a ratio of 1:1:1.

When the number of participants who have completed the 12-week follow up reached 120, interim analyses will be performed and the results will be evaluated by Independent Data Monitoring Committee experts to determine the recommended phase 3 dosage.

During the phase III stage, subjects were randomly assigned 1:1 to the "recommended phase 3 dosage + metformin" group and the "placebo + metformin" group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from 18 to 75;
2. Clinical diagnosed of Type 2 diabetes for at least 8 weeks ，receive metformin single treatment ；
3. During screening, HbA1c: 7.5% ≤ HbA1c ≤ 11% ，and before randomization 7.5% ≤ HbA1c ≤ 10.5%;
4. During screening and before randomization: FPG< 13.9 mmol/L； 5.18.5 kg/m2 ≤ BMI ≤ 35 kg/m2;

6. without birth plan and voluntarily take effective contraceptive measures; 7. fully understood the study, signed the informed consent；

Exclusion Criteria:

1. Diabetes other than Type 2;
2. Any dipeptidyl peptidase IV and / or glucagon-like peptide-1 （GLP-1）analogues were used within 3 months before screening;
3. Continuous use of insulin for more than 14 days in the previous year;
4. C-Peptide <0.3 nmol/L;
5. Diabetic ketoacidosis, diabetic lactic acidosis or hyperosmolar non ketonic diabetic coma occurred within 6 months before screening;
6. Unstable proliferative retinopathy or macular lesion, severe diabetic neuropathy, intermittent claudication or diabetic foot occurred within 6 months before screening;
7. Severe hypoglycemia occurred within 6 months before screening
8. Severe trauma infection or operation within one month before screening;
9. Blood donation or massive blood loss or transfusion within 3 months ;
10. Suspected active infection ;
11. Growth hormone therapy was performed within 6 months before screening;
12. Patients having received corticosteroid continuous ≥ 7 days through within 2 months ;
13. use any drugs or surgery with weight control effect within 2 months;
14. weight change of more than 5% within 3 months;
15. mean systolic pressure (SBP) ≥ 160mmhg and / or diastolic pressure （DBP） ≥ 90 mmHg at screening, or new/changed antihypertensive drugs or adjusted dosage of antihypertensive drugs within 4 weeks before screening or before induction period
16. with a history of severe cardiovascular disease, high risk of stroke/stroke within 6 months before screening;
17. with a history of acute or chronic pancreatitis, symptomatic gallbladder , pancreatic injury and other risk factors for pancreatitis, or with blood amylase and/or blood lipase ≥1.5 times the upper limit of normal (ULN) at the time of screening or before randomization;
18. Calcitonin level ≥50 ng/L (pg/mL) during screening;
19. with a history of medullary thyroid cancer, multiple endocrine neoplasm (Men) 2A or 2B syndrome, or related family history;
20. with clinically significant abnormal gastric emptying , severe chronic gastrointestinal diseases , long-term use of drugs that have a direct impact on gastrointestinal peristalsis , or having undergone gastrointestinal surgery within 6 months before screening, are not suitable to participate in this clinical study according to the evaluation of the researchers;
21. suffering from hematological diseases or any disease causing hemolysis or erythrocyte instability ;
22. Uncontrolled hyperthyroidism or hypothyroidism;
23. with hemoglobinopathy that may affect the determination of HbA1c levels;
24. HBsAg, Hepatitis C antibody, HIV-Ab, Treponema pallidum antibody or Corona Virus Disease 2019 nucleic acid tested positive;
25. serious mental illness;
26. drinking more than 14 standard units weekly within 6 months before screening ;
27. a history of organ transplantation or other acquired or congenital immune system diseases;
28. allergic to the active ingredients (GLP-1 and GLP-1 analogues) of the study drug;
29. clear contraindications for the use of metformin;
30. clear contraindications for Empagliflozin；
31. Any of the following conditions: the pacemaker was installed when screened; no pacemaker was installed, but 12 lead ECG showed degree II or III atrioventricular block, long QT syndrome or QTc interval ≥ 450ms ; Patients with New York Heart Function Classification III or IV; Or other abnormal cardiac function with clinical significance that is not suitable for clinical research judged by researchers;
32. acute or chronic hepatitis, or whose laboratory examination indexes meet one of the following criteria at the time of screening or before randomization : alanine aminotransferase (ALT) level ≥ 2.5 fold ULN, aspartate aminotransferase (AST) ≥ 2.5 fold ULN, fasting triglyceride (TG) > 5.7 mmol/L or 500 mg/dl; the glomerular filtration rate (EGFR) < 60 ml/min/1.73 square meters was calculated by CKD-EPI (epi - (SCR)) formula;
33. participated in clinical trials of other drugs or devices within 3 months before screening;
34. Medication compliance in the metformin dosage stable period was < 80% or > 120%;
35. Supaglutide placebo injection compliance during the induction period was <75% or>125%, or metformin compliance <80% or >120%;
36. Any other situation that researchers think may affect the patients' informed consent or compliance with the trial protocol;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-13 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  The change in mean HbA1c concentrations (%)from baseline with Supaglutide versus placebo

SECONDARY OUTCOMES:
fasting plasma glucose | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in fasting plasma glucose (mmol/L) relative to baseline
HbA1c<7.0% and <6.5% | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  The proportion of participants who achieved HbA1c target (HbA1c<7.0% and <6.5% Patient percentage)
Fasting insulin | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Fasting insulin changes（pmol/L) relative to baseline
fasting C-peptide | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Fasting C-peptide changes (nmol/L) relative to baseline
fasting glucagon | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  fasting glucagon changes (pg/ml) relative to baseline
Area under the curve of blood glucose | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Area under the curve of blood glucose (AUC0-120min,mmol/L) during the multi-maneuvering target tracking
Area under the curve of insulin | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Area under the curve of insulin (AUC0-120min,pmol/L) during the MMTT
Area under the curve of C-peptide | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Area under the curve of C-peptide (AUC0-120min,nmol/L) during the MMTT
Total cholesterol | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in total cholesterol (mmol/L) relative to baseline
low density lipoprotein | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in low density lipoprotein (mmol/L) relative to baseline
High density lipoprotein | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in high density lipoprotein (mmol/L) relative to baseline
triglyceride | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Changes in triglyceride(mmol/L) relative to baseline
weight | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Weight change from baseline(kg)
salvage treatment | 12 weeks for phase IIb; 24weeks and 52 weeks for phase III
  Percentage of subjects receiving salvage treatment(%)

CONTACTS AND LOCATIONS:
Overall Officials: Weiping Jia, M.D,Ph.D, Principal Investigator — Shanghai 6th People's Hospital
Locations (61):
- China (61):
  - Beijing Boai Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Emergency General Hospital, Beijing
  - Cangzhou Central Hospital, Cangzhou
  - Cangzhou Hospital of Integrated TCM-WM Hebei, Cangzhou
  - The Second Hospital of Jilin University, Changchun
  - First People's Hospital of Changde, Changde
  - Changsha Hopital Affiliated to Hunan University, Changsha
  - The Fourth Hospital of Changsha, Changsha
  - Chengdu Fifth People's Hospital, Chengdu
  - Chenzhou First People's Hospital, Chenzhou
  - Chongqing Ninth People's Hospital, Chongqing
  - Dalian Municipal Central Hospital, Dalian
  - Daqing People's Hospital, Daqing
  - Jilin Guowen Hospital, Gongzhuling
  - Handan First Hospital, Handan
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Heze Municipal Hospital, Heze
  - Huai'an First People's Hospital, Huai'an
  - Huai'an Second People's Hospital, Huai'an
  - Huizhou Central Hospital, Huizhou
  - Jilin People's Hospital, Jilin
  - Jinan Central Hospital Affiliated to Shandong First Medical University, Jinan
  - Jincheng General Hospital, Jincheng
  - Jingzhou Central Hospital, Jingzhou
  - The Second Affiliated Hospital of Kunming Medical University, Kunming
  - The Second People's Hospital of Lianyungang, Lianyungang
  - Linfen People's Hospital, Linfen
  - First People's Hospital of Tancheng, Linyi
  - Liuzhou People's Hospital, Liuchow
  - The First Affiliated Hospital of Henan University, Luoyang
  - Meihekou Central Hospital, Meihekou
  - Jiangxi Provincial People's Hospital, Nanchang
  - Nanjing First Hospital, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - Sir Run Run Hospital of Nanjing Medical University, Nanjing
  - Nanyang First People's Hospital, Nanyang
  - Nanyang Second General Hospital, Nanyang
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang
  - Puyang Oilfield General Hospital, Pujiang
  - The First Hospital of Qinhuangdao, Qinhuangdao
  - The First Hospital of Qiqihar, Qiqihar
  - Changhai Hospital, Shanghai
  - Huadong Hospital, Shanghai
  - Shanghai Pudong New Area People's Hospital, Shanghai
  - Shanghai Sixth People's Hospital Affiliated to Shanghai JiaoTong University, Shanghai
  - Shanghai Tongren Hospital, Shanghai
  - Siping Central Hospital, Siping
  - Second Hospital of Shanxi Medical University, Taiyuan
  - The Second Affiliated Hospital of Shandong First Medical University, Tanan
  - The Second Hospital of Tanjin Medical University, Tianjin
  - Tianjin Medical University General Hospital, Tianjing
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Jiangyin People's Hospital, Wuxi
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Xuzhou Cancer Hospital, Xuzhou
  - The Second People's Hospital of Yibin, Yibin
  - Yichun People's Hospital, Yichun
  - Yiyang Central Hospital, Yiyang
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou
  - First People's Hospital of Zunyi, Zunyi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Q, Jiang F, Xu Y, Lei Y, Zhang L, Sun X. Exposure-Response Analysis of Efsubaglutide Alfa in Patients with Type 2 Diabetes Treated with Metformin. Clin Pharmacokinet. 2025 Dec;64(12):1799-1809. doi: 10.1007/s40262-025-01569-2. Epub 2025 Sep 24. PMID 40991141
- [Derived] Lou YR, Xu YL, Xiong Y, Deng C, Wang Q. Population Pharmacokinetics of Efsubaglutide Alfa in Healthy Subjects and Subjects with Type 2 Diabetes. Clin Pharmacokinet. 2025 Apr;64(4):533-552. doi: 10.1007/s40262-025-01475-7. Epub 2025 Feb 17. PMID 39961992